CLINICAL TRIAL: NCT05785013
Title: The Impact of Preoperative Supplementation of Zinc on Post-operative Outcomes in Children Undergoing Elective Surgery for Hirsch Sprung Disease
Brief Title: The Impact of Preoperative Supplementation of Zinc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hoda Atef Abdelsattar Ibrahim, Lecturer of Pediatrics, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MS 277-2022
Record Dates: First submitted 2023-03-02; First posted 2023-03-27 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Surgery; Nutrition Disorders
MeSH Terms: conditions — Nutrition Disorders | interventions — Zinc

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional (Experimental): 25 children diagnosed with Hirschsprung disease and planned for elective surgery will be supplemented with Zinc 7 days before the operation . Outcomes will be evaluated thorugh measuring the hospital length stay. Other parameters including inflammatory markers as CRP , CRP /albumin ratio and development of postoperative complications will be assesed and compared between cases and controls
  Interventions: Dietary Supplement: Zinc
- Control (No Intervention): 25 children diagnosed with Hirschsprung disease and planned for elective surgery will recieve the standard care provided for the cases and will not be supplemented with Zinc . Outcomes will be evaluated thorugh measuring the hospital length. Other parameters including inflammatory markers as CRP , CRP /albumin ratio and development of postoperative complications will be assesed and compared between cases and controls

INTERVENTIONS:
Dietary Supplement: Zinc — Zinc Supplementation
  Arms: Interventional

SUMMARY:
1. Pre operative anthropometric assessment including : weight in kg, height/length and BMI
2. Pre operative Zinc supplementation (dose according to the age) for 7 days preoperatively for cases
3. Postoperative data collection

DETAILED DESCRIPTION:
Postoperative data collection :

* Length of hospital stay
* Complication and sorting of them
* Lab withdrawal of inflammatory markers on 2-3 day postoperatively

ELIGIBILITY:
Inclusion Criteria:

1. All children patients with Hirschsprung disease admitted for surgical intervention with different ( age , sex )
2. Type of surgery : transanal pull through
3. Whose parents or caregivers approve for the participation in the study

Exclusion Criteria:

1. Patients with emergency situations
2. Whose parents or caregivers will not apply for the participation in the study

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-02 (Actual)

PRIMARY OUTCOMES:
The effect of preoerative Zinc supplementation on the hospital length stay in children operated for Hirschsprung's disease | zinc supplemenation for one week
  Children oprated for elective surgery for Hirschsprung's disease will be supplemented with zinc seven days before surgery and postoperative data as the duration of hospital length stay in hours will be meausred in both the cases and control groups and comapred.

CONTACTS AND LOCATIONS:
Locations (1):
- Hoda Atef Abdelsattar Ibrahim, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Anonoymus data can be reproduced